CLINICAL TRIAL: NCT05673668
Title: Clinical Mechanism of Endovascular Denervation (EDN) for the Treatment of Type 2 Diabetes
Brief Title: Endovascular Denervation (EDN) for the Treatment of Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Clinical Professor, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDN-T2DM
Record Dates: First submitted 2022-11-28; First posted 2023-01-06 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Type 2 Diabetes Mellitus; Endovascular denervation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The endovascular denervation (EDN) group (Experimental): Receive endovascular denervation (EDN) treatment
  Interventions: Device: Endovascular Denervation System (Netrod)

INTERVENTIONS:
Device: Endovascular Denervation System (Netrod) — The Netrod system is a percutaneous, catheter- based device which uses radiofrequency energy to denervate the sympathetic nerves surrounding the arteries

SUMMARY:
This is a prospective, single-center, single-arm, self-controlled study to evaluate the effects of endovascular denervation (EDN) on insulin secretory function and insulin sensitivity in the treatment of type 2 diabetes mellitus (T2DM) .

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, self-controlled study. Patients with diagnosed T2DM and poor glycemic control (i.e.. glycated hemoglobin A1c (HbA1c) between 7.5% and 10.5% despite one to three oral antidiabetic drugs (OAD) and/or insulin on the basis of metformin. All included subjects will accept EDN treatment and were followed up at 7, 30 days and 3, 6, 12 months. The primary objectives were evaluate the effects of EDN on insulin secretory function and insulin sensitivity in the treatment of T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with age of #18 years old and#75 years old (both ends included)
2. Subject (or legal guardian) understands the requirements and treatment of this clinical trial and agrees to and is able to complete the trial
3. Diagnosed with T2DM for ≤15 years (according to WHO criteria)
4. On the basis of metformin (daily dose ≥1000mg), using a combination of 1-3 OADs for more than last 3 months, with or without insulin (dose not limited). Defined OADs were: sulfonylureas/ glienides, thiazolidinediones and α-glycosidase inhibitors
5. Glycosylated hemoglobin (HbA1c) levels between 7.5% and 10.5% (based on baseline tests)
6. Body mass index (BMI) ≥ 18 and ≤40kg/m2

Exclusion Criteria:

1. T1DM or any secondary diabetes
2. History of aortic disease (such as aortic aneurysm or aortic dissection) or aortic surgery (including celiac artery dissection)
3. Baseline CTA examination revealed aortic aneurysm or aortic dissection, or abnormal anatomical structure of hepatic artery and its branches, or other vascular structure/status abnormalities (such as severe tortuosity or narrowing of the artery, endovascular thrombosis or unstable plaque, etc.) that were not suitable for endovascular denervation as determined by the researcher
4. More than 2 self-reported or documented events of severe hypoglycemia (defined as hypoglycemia with severe cognitive impairment requiring assistance) within the past 6 months
5. Patients who had a major cardiovascular and cerebrovascular event (MACCE), major surgery, severe infection, gastrointestinal bleeding, and acute pancreatitis in the past 6 months
6. Severe autonomic neuropathy (postural hypotension, etc.)
7. Severe liver insufficiency (ALT and/or AST above 3 times the normal upper limit or serum total bilirubin above 2 times the normal upper limit), renal insufficiency (eGFR < 60mL/ min/1.73m2). eGFR calculation formula is shown in Note e of Table 4.3 Data collection table.), chronic pancreatitis, cocoagulation disorder (PT, APTT or INR higher than 2 times of the normal upper limit; Platelet count < 80×109/L or ≥ 700×109/L) and malignant tumors
8. Suffering from mental illness and unable to cooperate
9. Pregnant
10. There were conditions that the researchers determined will affect the safety of the subjects or interfere with the evaluation of the test results
11. Patients not eligible for MRI (e.g. paramagnetic metal implants, claustrophobia, etc.)
12. Participating in or currently participating in other clinical studies within 3 months prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes of islet secretory function (HOMA-β) | From baseline to 6 months
  Changes of islet secretory function (HOMA-β, HOMA-IR) from baseline at 6 months post procedure

SECONDARY OUTCOMES:
Incidence of device or procedure-related major adverse events | From baseline to 12 months post procedure
  Incidence of device or procedure-related major adverse events from baseline to 12 months post procedure
Changes in Hba1c | From baseline to 12 months post procedure
  Changes in Hba1c from baseline at 12 months post procedure
Changes in the time in range (TIR) over 14 days of glucose | From baseline to 12 months post procedure
  Changes in the time in range (TIR) over 14 days of using continuous glucose monitoring at 12 months post procedure
Changes in the area under OGTT insulin release curve | From baseline to 12 months post procedure
  Change in the area under OGTT insulin release curve from base line to 12 months post procedure
Changes in the area under OGTT C-peptide release curve | From baseline to 12 months post procedure
  Changes in the area under OGTT C-peptide release curve from base line to 12 months post procedure
Changes in liver fat content | From baseline to 6 months post procedure
  Changes in liver fat content from baseline at 6 months post procedure
Changes in liver function | From baseline to 6 months post procedure
  Changes of liver function (ALT, AST, GGT, ALP) from baseline at 6 months post procedure
Changes in blood lipids | From baseline to 12 months post procedure
  Changes in blood lipid as indicated by triglycerides, total cholesterol, HDL cholesterol and LDL cholesterol from baseline at 12 months post procedure
Changes in the gastric emptying | From baseline to 12 months post procedure
  Changes in the gastric emptying as indicated by 13C-acetate breath test from baseline at 12 months post procedure
Changes in insulin sensitivity | From baseline to 6 months post procedure
  Changes in insulin sensitivity as indicated by glucose infusion rate and M value in hyperinsulinemic-euglycemic clamp from baseline at 6 months post procedure
Changes in metabolic-related hormones | From baseline to 6 months post procedure
  Changes in metabolic-related hormones including glucagon, pancreatic polypeptide, glucagon-like peptide-1, gastric inhibitory polypeptide, neuropeptide Y, peptide YY, ghrelin, adiponectin and leptin
Changes in plasma cytokines | From baseline to 6 months post procedure
  Changes in plasma cytokines including IFN-γ、IL-1β、IL-2、IL-4、IL-6、IL-10、IL-12p70、IL-17A、TNF-α、IL-13、IL-15、MCP-1、FGF21/23 and BDNF from baseline at 6 months post procedure
Changes in blood and fecal metabolome | From baseline to 6 months post procedure
  Changes in blood and fecal metabolome (Using liquid-mass combination (LC - MS) method) from baseline at 6 months post procedure
Changes in fecal microbiota | From baseline to 6 months post procedure
  Changes in fecal microbiota (Using liquid-mass combination (LC - MS) method assess fecal 16S-rRNA sequencing and non-targeted metabolomics) from baseline at 6 months post procedure
Change of sympathetic nervous system activity | From baseline to 6 months post procedure
  Change of sympathetic nervous system activity (cardiac strain capacity was evaluated by autonomic nervous function and Cardiopulmonary resonance assesses sympathetic nervous system excitability) from baseline at 6 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China